CLINICAL TRIAL: NCT02455180
Title: Pharmacokinetics of Two Different High-dose Regimens of Intravenous Vitamin C in Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, H.M. Oudemans-van Straaten, MD, PhD, Intensivist, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL50578.029.14; 2014-003680-38 (EudraCT Number)
Record Dates: First submitted 2015-05-21; First posted 2015-05-27 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Multiple Organ Failure; Sepsis; Systemic Inflammatory Response Syndrome; Trauma
Keywords: Critical Care
MeSH Terms: conditions — Multiple Organ Failure; Sepsis; Systemic Inflammatory Response Syndrome; Wounds and Injuries | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 4x 1 gram bolus (q12H) dosage regimen (Experimental): 1 gram of intravenous Vitamin C (ascorbic acid) is given 4 times at 12 hour intervals (total dose 4 grams).
  Interventions: Drug: Ascorbic Acid
- 4x 5 grams bolus (q12H) dosage regimen (Experimental): 5 grams of intravenous Vitamin C (ascorbic acid) is given 4 times at 12 hour intervals (total dose 20 grams).
  Interventions: Drug: Ascorbic Acid
- 4 gram continuous dosage regimen (Experimental): 1 gram per 12 hours of intravenous Vitamin C (ascorbic acid) is given continuously for 48 hours
  Interventions: Drug: Ascorbic Acid
- 20 gram continuous dosage regimen (Experimental): 5 gram per 12 hours of intravenous Vitamin C (ascorbic acid) is given continuously for 48 hours
  Interventions: Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Ascorbic Acid — Patients receive vitamin C 4 times in either high (5g) or moderate (1g) dose. Vitamin C will be administered intravenously (ascorbinezuur CF 100 mg/ml, Centrafarm BV, Etten Leur, Netherlands) in 50ml of NaCl 0.9%, infused over 30 minutes.
  Other Names: Vitamin C

SUMMARY:
The purpose of this study is to determine the pharmacokinetic properties of two different dosage regimens of intravenous vitamin C in patients admitted to the Intensive Care Unit with life-threatening illness.

DETAILED DESCRIPTION:
Rationale:

Critically ill patients with trauma or sepsis exhibit a high degree of vitamin C deficiency at ICU admission and vitamin C plasma concentrations decrease even more during the first three days of admission. Vitamin C is a natural anti-oxidant and crucial for endothelial and organ protection

Objective:

To determine the pharmacokinetics of two high dose regimens of intravenous vitamin C in critically ill patients, in particular the attained plasma concentration and the fraction retained in the body and excreted in urine.

Study design:

Prospective randomized controlled pharmacokinetic intervention study

Study population:

Adult critically ill patients admitted to the ICU of the VU University Medical Center, Amsterdam, with sepsis or SIRS after major surgery or trauma with a non-neurological sequential organ failure (SOFA) score >6 and an expected length of ICU stay of >96 hours.

Intervention (if applicable):

Patients will receive either 2 or 10 gram/day vitamin C intravenously twice daily for two days in bolus or continuous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis or Systemic Inflammatory Response Syndrome (SIRS) after major surgery or trauma;
* Non-neurological sequential organ failure assessment (SOFA) score >6;
* Expected length of ICU stay > 96 hours;
* Written proxy consent by legal representative.

Exclusion Criteria:

* Admission after out of hospital cardiac arrest
* Prior use of supplemental vitamin C in the week before
* Major bleeding
* Pre-existent renal insufficiency defined as an eGFR of < 30 ml/min/1.73 m2 (stadium 4-5)
* Expected need for renal replacement therapy within 48 hours
* Known glucose 6-phosphate dehydrogenase deficiency
* History of urolithiasis or oxalate nephropathy
* Previous use of prolonged high dose vitamin C supplements
* Hemochromatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Vitamin C plasma concentration | Baseline (before intervention), thereafter at 1, 2, 4, 8, 12, 24, 36, 48, 72, 96 hours after first intervention
Vitamin C excreted in urine | 0-12hours after first intervention; 36-48 hours after first intervention

SECONDARY OUTCOMES:
Oxalate excretion in urine | 0-12hours after first intervention; 36-48 hours after first intervention
F2-isoprostanes (oxidative damage biomarker) | 0, 24 and 72 hours after first intervention
CellROX (reactive oxygen species activity in leukocytes) | 0 and 24 hours after first intervention
Vasopressor requirements (noradrenalin dose) | 0, 12, 24, 48, 72 and 96 hours after first intervention
Renal resistive index (ultrasonography) | 0, 4, 24, 72 hours after first intervention
Serum creatinine and creatinine clearance | 0, 24, 48, 72, 95 after first intervention
Sequential Organ Failure Assessment (SOFA) score | 0, 24, 48, 72, 95 after first intervention

CONTACTS AND LOCATIONS:
Overall Officials: H.M. Oudemans-van Straaten, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] de Grooth HJ, Manubulu-Choo WP, Zandvliet AS, Spoelstra-de Man AME, Girbes AR, Swart EL, Oudemans-van Straaten HM. Vitamin C Pharmacokinetics in Critically Ill Patients: A Randomized Trial of Four IV Regimens. Chest. 2018 Jun;153(6):1368-1377. doi: 10.1016/j.chest.2018.02.025. Epub 2018 Mar 6. PMID 29522710